CLINICAL TRIAL: NCT01669915
Title: A Large Randomized Trial of Vitamin D, Omega-3 Fatty Acids and Cognitive Decline
Acronym: VITAL-Cog
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jae Hee Kang, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2010P-000769; R01AG036755 (NIH)
Record Dates: First submitted 2012-08-17; First posted 2012-08-21 (Estimated); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-03

CONDITIONS: Cognitive Decline
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cholecalciferol; Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ACTIVE Vitamin D + ACTIVE Omega-3 Fatty Acids (Active Comparator): ACTIVE Vitamin D = Vitamin D3, one 2000 IU capsule/day; ACTIVE Omega-3 Fatty Acids = Omacor, one 1-gram capsule/day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Interventions: Dietary Supplement: vitamin D3; Drug: omega-3 fatty acids (fish oil)
- ACTIVE Vitamin D + PLACEBO Omega-3 Fatty Acids (Active Comparator): ACTIVE Vitamin D = Vitamin D3, one 2000 IU capsule/day; PLACEBO Omega-3 Fatty Acids, one capsule/day
  Interventions: Dietary Supplement: vitamin D3; Dietary Supplement: Fish oil placebo
- PLACEBO Vitamin D + ACTIVE Omega-3 Fatty Acids (Active Comparator): PLACEBO Vitamin D, one capsule/day; ACTIVE Omega-3 Fatty Acids = Omacor, one 1-gram capsule/day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Interventions: Drug: omega-3 fatty acids (fish oil); Dietary Supplement: Vitamin D3 placebo
- PLACEBO Vitamin D + PLACEBO Omega-3 Fatty Acids (Placebo Comparator): PLACEBO Vitamin D, one capsule/day; PLACEBO Omega-3 Fatty Acids, one capsule/day
  Interventions: Dietary Supplement: Vitamin D3 placebo; Dietary Supplement: Fish oil placebo

INTERVENTIONS:
Dietary Supplement: vitamin D3 — Vitamin D3 (cholecalciferol), 2000 IU per day
  Other Names: cholecalciferol
  Arms: ACTIVE Vitamin D + ACTIVE Omega-3 Fatty Acids; ACTIVE Vitamin D + PLACEBO Omega-3 Fatty Acids
Drug: omega-3 fatty acids (fish oil) — Omacor, 1 capsule per day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
  Arms: ACTIVE Vitamin D + ACTIVE Omega-3 Fatty Acids; PLACEBO Vitamin D + ACTIVE Omega-3 Fatty Acids
Dietary Supplement: Vitamin D3 placebo — Vitamin D placebo
  Arms: PLACEBO Vitamin D + ACTIVE Omega-3 Fatty Acids; PLACEBO Vitamin D + PLACEBO Omega-3 Fatty Acids
Dietary Supplement: Fish oil placebo — Fish oil placebo
  Arms: ACTIVE Vitamin D + PLACEBO Omega-3 Fatty Acids; PLACEBO Vitamin D + PLACEBO Omega-3 Fatty Acids

SUMMARY:
The VITamin D and OmegA-3 TriaL (VITAL; NCT 01169259) is an ongoing randomized clinical trial in 25,875 U.S. men and women investigating whether taking daily dietary supplements of vitamin D3 (2000 IU) or omega-3 fatty acids (Omacor® fish oil, 1 gram) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses. This ancillary study is being conducted among participants in VITAL and will examine whether vitamin D or fish oil is associated with cognitive decline in 3000 older participants of VITAL.

DETAILED DESCRIPTION:
Primary aim of annual rate of cognitive decline. Secondary aims will be addressed in sub-set of participants: 1) among participants, African-American race (African-Americans have high risk of Vitamin D deficiency) modifies effects of vitamin D3 supplementation on cognitive decline; 2) among a subset of participants, baseline plasma levels of vitamin D and omega-3 fatty acids modify agent effects.

ELIGIBILITY:
Participants in VITAL (NCT 01169259) who meet the following criteria are eligible to participate in this ancillary study:

1. are aged 60 or more
2. have no hearing impairment
3. indicate a willingness on the run-in phase to participate in a cognitive sub-study.

Ages: 60 Years to 92 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3424 (Actual)
Dates: Start 2011-09-14 (Actual); Primary Completion 2016-06-08 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Kang JH, Vyas CM, Okereke OI, Ogata S, Albert M, Lee IM, D'Agostino D, Buring JE, Cook NR, Grodstein F, Manson JE. Effect of vitamin D on cognitive decline: results from two ancillary studies of the VITAL randomized trial. Sci Rep. 2021 Dec 1;11(1):23253. doi: 10.1038/s41598-021-02485-8. PMID 34853363
- See also: VITAL study website link — http://www.vitalstudy.org

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this telephone interview ancillary study, participants (NCT01169259) who:1) were aged 60 or more; 2) had no hearing impairment; 3) were willing to participate in a cognitive sub-study (during run-in phase) were included.
Groups:
- TELEPHONE INTERVIEW ANCILLARY STUDY: ACTIVE Vitamin D + ACTIVE Omega-3 Fatty Acids: ACTIVE Vitamin D = Vitamin D3, one 2000 IU capsule/day; ACTIVE Omega-3 Fatty Acids = Omacor, one 1-gram capsule/day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
- TELEPHONE INTERVIEW ANCILLARY STUDY: ACTIVE Vitamin D + PLACEBO Omega-3 Fatty Acids: ACTIVE Vitamin D = Vitamin D3, one 2000 IU capsule/day; PLACEBO Omega-3 Fatty Acids, one capsule/day
- TELEPHONE INTERVIEW ANCILLARY STUDY: PLACEBO Vitamin D + ACTIVE Omega-3 Fatty Acids: PLACEBO Vitamin D, one capsule/day; ACTIVE Omega-3 Fatty Acids = Omacor, one 1-gram capsule/day. Each capsule of Omacor contains 840 milligrams of marine omega-3 fatty acids (465 mg of eicosapentaenoic acid [EPA] and 375 mg of docosahexaenoic acid [DHA]).
- TELEPHONE INTERVIEW ANCILLARY STUDY: PLACEBO Vitamin D + PLACEBO Omega-3 Fatty Acids: PLACEBO Vitamin D, one capsule/day; PLACEBO Omega-3 Fatty Acids, one capsule/day
Period: Overall Study
Arm/Group | TELEPHONE INTERVIEW ANCILLARY STUDY: ACTIVE Vitamin D + ACTIVE Omega-3 Fatty Acids | TELEPHONE INTERVIEW ANCILLARY STUDY: ACTIVE Vitamin D + PLACEBO Omega-3 Fatty Acids | TELEPHONE INTERVIEW ANCILLARY STUDY: PLACEBO Vitamin D + ACTIVE Omega-3 Fatty Acids | TELEPHONE INTERVIEW ANCILLARY STUDY: PLACEBO Vitamin D + PLACEBO Omega-3 Fatty Acids
Started | 844 | 866 | 855 | 859
Completed | 844 | 866 | 855 | 859
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TELEPHONE INTERVIEW ANCILLARY STUDY: ACTIVE Vitamin D + ACTIVE Omega-3 Fatty Acids | TELEPHONE INTERVIEW ANCILLARY STUDY: ACTIVE Vitamin D + PLACEBO Omega-3 Fatty Acids | TELEPHONE INTERVIEW ANCILLARY STUDY: PLACEBO Vitamin D + ACTIVE Omega-3 Fatty Acids | TELEPHONE INTERVIEW ANCILLARY STUDY: PLACEBO Vitamin D + PLACEBO Omega-3 Fatty Acids | Total
Number analyzed (Participants) | 844 | 866 | 855 | 859 | 3424
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 95 | 115 | 88 | 90 | 388
  >=65 years | 749 | 751 | 767 | 769 | 3036
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (6.0) | 70.8 (5.9) | 71.1 (6.0) | 70.7 (5.7) | 70.9 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 484 | 527 | 503 | 502 | 2016
  Male | 360 | 339 | 352 | 357 | 1408
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic white | 595 | 589 | 624 | 621 | 2429
  African American | 178 | 209 | 181 | 175 | 743
  Hispanic (not African American) | 12 | 19 | 13 | 17 | 61
  Asian/Pacific Islander | 16 | 9 | 8 | 8 | 41
  Native American/Alaskan Native | 20 | 14 | 14 | 25 | 73
  Other/unknown | 23 | 26 | 15 | 13 | 77
Region of Enrollment [Number; unit: participants]
  United States | 844 | 866 | 855 | 859 | 4218

OUTCOME MEASURES:

1. Primary Outcome: Change in Global Composite Score for Cognitive Decline
Description: We administered by telephone, eight cognitive tests (1.Telephone Interview of Cognitive Status (TICS); 2.Delayed recall of the TICS 10-word list; 3.East Boston Memory Test (EBMT); 4.Delayed recall of the EBMT; 5.Category fluency test (animal naming test); 6.Oral Trail Making Test (OTMT-Part A); 7. OTMT-Part B; 8.Digit span backwards). The primary endpoint was the change over time (last assessment score minus the baseline assessment score) in GLOBAL COMPOSITE SCORE (average of Z-scores of component tests); for both baseline and last assessment Z-scores, a mean Z-score of 0 represents the mean and the higher the Z-score, the better the overall cognitive performance across the tests. The primary endpoint was a difference of two Z-scores, so a value of 0 means no change over time, a positive value means an increase over time and a negative value means a decrease (or "decline") over time, for clinical significance, 1 year of aging is associated with a primary endpoint value of -0.004.
Time Frame: Change over two assessments (baseline, 2.8 years).
Measure: Mean (Standard Error); unit: Z-score
Groups:
- TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D: Vitamin D3, one 2000 IU capsule/day
- TELEPHONE INTERVIEW ANCILLARY STUDY: Vitamin D Placebo: Vitamin D placebo, one capsule/day
- TELEPHONE INTERVIEW ANCILLARY STUDY: Active Omega-3 Fatty Acids: Omacor, one 1-g capsule/day. Each capsule of Omacor contains 840 mg of marine omega-3 fatty acids (465 mg of EPA + 375 mg of DHA).
- TELEPHONE INTERVIEW ANCILLARY STUDY: Omega-3 Fatty Acids Placebo: Omega-3 fatty acids placebo, one capsule/day
Arm/Group | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D | TELEPHONE INTERVIEW ANCILLARY STUDY: Vitamin D Placebo | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Omega-3 Fatty Acids | TELEPHONE INTERVIEW ANCILLARY STUDY: Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 1710 | 1714 | 1699 | 1725
Z-score | -0.24 (0.01) | -0.25 (0.01) | -0.25 (0.01) | -0.24 (0.01)
Statistical Analysis 1: Comparison: TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D vs TELEPHONE INTERVIEW ANCILLARY STUDY: Vitamin D Placebo; The rates of cognitive decline over 2.8 years were compared in the two groups (rate in vitamin D active group minus the rate in placebo group). A mixed model included terms for the variables time since randomization, assignment to one arm, assignment to the other arm, sex, age, race/ethnicity, history of depression and the six interaction terms (products with time since randomization); Test type: Superiority; p = 0.31, Mixed Models Analysis; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.01 to 0.02]
Statistical Analysis 2: Comparison: TELEPHONE INTERVIEW ANCILLARY STUDY: Active Omega-3 Fatty Acids vs TELEPHONE INTERVIEW ANCILLARY STUDY: Omega-3 Fatty Acids Placebo; The rates of cognitive decline over 2.8 years were compared in the two groups (rate in omega-3 fatty acids active group minus the rate in placebo group). A mixed model included the variables, time since randomization, assignment to one arm, assignment to the other arm, sex, age, race/ethnicity, history of depression and the six interaction terms (products with time since randomization); Test type: Superiority; p = 0.14, Mixed Models Analysis; Mean Difference (Net) = -0.01, 95% CI 2-sided [-0.02 to 0.003]

2. Secondary Outcome: Change in Episodic Memory Score for Cognitive Decline
Description: The outcome measure was change over time (last assessment score minus the baseline assessment score) in the EPISODIC MEMORY SCORE combining z-scores of 4 tests: the immediate and delayed recalls of both the East Boston Memory Test (EBMT) and the Telephone Interview of Cognitive Status (TICS) 10-word list; for both baseline and last assessment Z-scores, a mean Z-score of 0 represents the mean and the higher the Z-score, the better the overall cognitive performance across the tests. The primary endpoint was a difference of two Z-scores, so a value of 0 means no change over time, a positive value means an increase over time and a negative value means a decrease (or "decline") over time, for clinical significance, 1 year of aging is associated with a primary endpoint value of -0.01.
Time Frame: Change over two assessments (baseline, 2.8 years)
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D | TELEPHONE INTERVIEW ANCILLARY STUDY: Vitamin D Placebo | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Omega-3 Fatty Acids | TELEPHONE INTERVIEW ANCILLARY STUDY: Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 1710 | 1714 | 1699 | 1725
Z-score | 0.00 (0.02) | -0.02 (0.02) | -0.03 (0.02) | 0.02 (0.02)
Statistical Analysis 1: Comparison: TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D vs TELEPHONE INTERVIEW ANCILLARY STUDY: Vitamin D Placebo; The rates of cognitive decline over 2.8 years were compared in the two groups (rate in vitamin D active group minus the rate in placebo group). A mixed model included the variables, time since randomization, assignment to one arm, assignment to the other arm, sex, age, race/ethnicity, history of depression and the six interaction terms (products with time since randomization); Test type: Superiority; p = 0.49, Mixed Models Analysis — Given the 3 secondary analyses, the p-value threshold was 0.0167 (=Bonferroni correction of 0.05/3=0.0167); Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.01 to 0.03]
Statistical Analysis 2: Comparison: TELEPHONE INTERVIEW ANCILLARY STUDY: Active Omega-3 Fatty Acids vs TELEPHONE INTERVIEW ANCILLARY STUDY: Omega-3 Fatty Acids Placebo; The rates of cognitive decline over 2.8 years were compared in the two groups (rate in omega-3 active group minus the rate in placebo group). A mixed model included the variables, time since randomization, assignment to one arm, assignment to the other arm, sex, age, race/ethnicity, history of depression and the six interaction terms (products with time since randomization); Test type: Superiority; p = 0.03, Mixed Models Analysis — Given the 3 secondary analyses, the p-value threshold was 0.0167 (=Bonferroni correction of 0.05/3=0.0167); Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.04 to -0.002]

3. Secondary Outcome: Change in Executive Function Score for Cognitive Decline
Description: The outcome measure is change over time (last assessment score minus the baseline assessment score) in the EXECUTIVE FUNCTION SCORE combining z-scores of 4 tests: category fluency (animal naming), digit span backwards, and Oral Trails Making Test (OTMT)-Part A and OTMT-Part B; for both baseline and last assessment Z-scores, a mean Z-score of 0 represents the mean and the higher the Z-score, the better the overall cognitive performance across the tests. The primary endpoint was a difference of two Z-scores, so a value of 0 means no change over time, a positive value means an increase over time and a negative value means a decrease (or "decline") over time, for clinical significance, 1 year of aging is associated with a primary endpoint value of +0.006.
Time Frame: Change over two assessments (baseline, 2.8 years)
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D | TELEPHONE INTERVIEW ANCILLARY STUDY: Vitamin D Placebo | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Omega-3 Fatty Acids | TELEPHONE INTERVIEW ANCILLARY STUDY: Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 1710 | 1714 | 1699 | 1725
Z-score | -0.48 (0.02) | -0.48 (0.02) | -0.47 (0.02) | -0.49 (0.02)
Statistical Analysis 1: Comparison: TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D vs TELEPHONE INTERVIEW ANCILLARY STUDY: Vitamin D Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.23, Mixed Models Analysis — Given the 3 secondary analyses, the p-value threshold was 0.0167 (=Bonferroni correction of 0.05/3=0.0167); Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.01 to 0.02]
Statistical Analysis 2: Comparison: TELEPHONE INTERVIEW ANCILLARY STUDY: Active Omega-3 Fatty Acids vs TELEPHONE INTERVIEW ANCILLARY STUDY: Omega-3 Fatty Acids Placebo; The rates of cognitive decline over 2.8 years were compared in the two groups (rate in omega-3 active group minus the rate in placebo group). A mixed model included terms for the variables time since randomization, assignment to one arm, assignment to the other arm, sex, age, race/ethnicity, history of depression and the six interaction terms (products with time since randomization); Test type: Superiority; p = 0.68, Mixed Models Analysis — Given the 3 secondary analyses, the p-value threshold was 0.0167 (=Bonferroni correction of 0.05/3=0.0167); Mean Difference (Net) = 0.003, 95% CI 2-sided [-0.01 to 0.02]

4. Secondary Outcome: Change in Telephone Interview of Cognitive Status (TICS) for Cognitive Decline.
Description: Change over time (last assessment score minus the baseline assessment score) on the TICS (0-41 points), a measure of general cognition. A higher value on the TICS represents better cognitive performance; for clinical significance, 1 year of aging is associated with a primary endpoint value of -0.05
Time Frame: Change over two assessments (baseline, 2.8 years)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D | TELEPHONE INTERVIEW ANCILLARY STUDY: Vitamin D Placebo | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Omega-3 Fatty Acids | TELEPHONE INTERVIEW ANCILLARY STUDY: Omega-3 Fatty Acids Placebo
Number analyzed (Participants) | 1710 | 1714 | 1699 | 1725
score on a scale | 0.12 (0.07) | 0.07 (0.07) | 0.005 (0.07) | 0.18 (0.07)
Statistical Analysis 1: Comparison: TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D vs TELEPHONE INTERVIEW ANCILLARY STUDY: Vitamin D Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.46, Mixed Models Analysis — Given the 3 secondary analyses, the p-value threshold was 0.0167 (=Bonferroni correction of 0.05/3=0.0167); Mean Difference (Net) = 0.03, 95% CI 2-sided [-0.04 to 0.09]
Statistical Analysis 2: Comparison: TELEPHONE INTERVIEW ANCILLARY STUDY: Active Omega-3 Fatty Acids vs TELEPHONE INTERVIEW ANCILLARY STUDY: Omega-3 Fatty Acids Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.003, Mixed Models Analysis — Given the 3 secondary analyses, the p-value threshold was 0.0167 (=Bonferroni correction of 0.05/3=0.0167); Mean Difference (Net) = -0.10, 95% CI 2-sided [-0.17 to -0.04]

ADVERSE EVENTS:
Groups:
- TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D/Active Omega-3 Fatty Acids: Vitamin D3 (one 2000 IU capsule/day) + Omacor, one 1-g capsule/day. Each capsule of Omacor contains 840 mg of marine omega-3 fatty acids (465 mg of EPA + 375 mg of DHA).
- TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D/Placebo Omega-3 Fatty Acids: Vitamin D3, one 2000 IU capsule/day + Omega-3 fatty acids placebo, one capsule/day
- TELEPHONE INTERVIEW ANCILLARY STUDY: Placebo Vitamin D/Active Omega-3 Fatty Acids: Vitamin D placebo, one capsule/day + Omacor, one 1-g capsule/day. Each capsule of Omacor contains 840 mg of marine omega-3 fatty acids (465 mg of EPA + 375 mg of DHA).
- TELEPHONE INTERVIEW ANCILLARY STUDY: Placebo Vitamin D/Placebo Omega-3 Fatty Acids: Vitamin D placebo, one capsule/day + Omega-3 fatty acids placebo, one capsule/day
Arm/Group | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D | TELEPHONE INTERVIEW ANCILLARY STUDY: Vitamin D Placebo | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Omega-3 Fatty Acids | TELEPHONE INTERVIEW ANCILLARY STUDY: Omega-3 Fatty Acids Placebo | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D/Active Omega-3 Fatty Acids | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D/Placebo Omega-3 Fatty Acids | TELEPHONE INTERVIEW ANCILLARY STUDY: Placebo Vitamin D/Active Omega-3 Fatty Acids | TELEPHONE INTERVIEW ANCILLARY STUDY: Placebo Vitamin D/Placebo Omega-3 Fatty Acids
All-Cause Mortality (participants affected / at risk) | 41/1710 | 26/1714 | 42/1699 | 25/1725 | 26/844 | 15/866 | 16/855 | 10/859
Serious Adverse Events (participants affected / at risk) | 138/1710 | 117/1714 | 134/1699 | 121/1725 | 74/844 | 64/866 | 60/855 | 57/859
Other Adverse Events (participants affected / at risk) | 1259/1710 | 1236/1714 | 1220/1699 | 1275/1725 | 600/844 | 659/866 | 620/855 | 616/859
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D (N=1710) | TELEPHONE INTERVIEW ANCILLARY STUDY: Vitamin D Placebo (N=1714) | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Omega-3 Fatty Acids (N=1699) | TELEPHONE INTERVIEW ANCILLARY STUDY: Omega-3 Fatty Acids Placebo (N=1725) | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D/Active Omega-3 Fatty Acids (N=844) | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D/Placebo Omega-3 Fatty Acids (N=866) | TELEPHONE INTERVIEW ANCILLARY STUDY: Placebo Vitamin D/Active Omega-3 Fatty Acids (N=855) | TELEPHONE INTERVIEW ANCILLARY STUDY: Placebo Vitamin D/Placebo Omega-3 Fatty Acids (N=859)
Death (General disorders) | 41 (41) | 26 (26) | 42 (42) | 25 (25) | 26 (26) | 15 (15) | 16 (16) | 10 (10) — Death
Cancer (General disorders) | 62 (62) | 51 (51) | 54 (54) | 59 (59) | 30 (30) | 32 (32) | 24 (24) | 27 (27) — Cancer
Gastrointestinal bleeding (Gastrointestinal disorders) | 25 (25) | 33 (33) | 34 (34) | 24 (24) | 14 (14) | 11 (11) | 20 (20) | 13 (13) — Gastrointestinal bleeding
Hypercalcemia (Blood and lymphatic system disorders) | 12 (12) | 5 (5) | 10 (10) | 7 (7) | 8 (8) | 4 (4) | 2 (2) | 3 (3)
Major cardiovascular event (Cardiac disorders) | 37 (37) | 22 (22) | 35 (35) | 24 (24) | 24 (24) | 13 (13) | 11 (11) | 11 (11)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D (N=1710) | TELEPHONE INTERVIEW ANCILLARY STUDY: Vitamin D Placebo (N=1714) | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Omega-3 Fatty Acids (N=1699) | TELEPHONE INTERVIEW ANCILLARY STUDY: Omega-3 Fatty Acids Placebo (N=1725) | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D/Active Omega-3 Fatty Acids (N=844) | TELEPHONE INTERVIEW ANCILLARY STUDY: Active Vitamin D/Placebo Omega-3 Fatty Acids (N=866) | TELEPHONE INTERVIEW ANCILLARY STUDY: Placebo Vitamin D/Active Omega-3 Fatty Acids (N=855) | TELEPHONE INTERVIEW ANCILLARY STUDY: Placebo Vitamin D/Placebo Omega-3 Fatty Acids (N=859)
Easy bruising (Blood and lymphatic system disorders) | 432 (432) | 411 (411) | 429 (429) | 414 (414) | 213 (213) | 219 (219) | 216 (216) | 195 (195)
Frequent nosebleeds (Blood and lymphatic system disorders) | 43 (43) | 56 (56) | 50 (50) | 49 (49) | 23 (23) | 20 (20) | 27 (27) | 29 (29)
Blood in urine (Blood and lymphatic system disorders) | 79 (79) | 81 (81) | 88 (88) | 72 (72) | 41 (41) | 38 (38) | 47 (47) | 34 (34)
Parathyroid condition (Endocrine disorders) | 5 (5) | 6 (6) | 6 (6) | 5 (5) | 3 (3) | 2 (2) | 3 (3) | 3 (3)
Stomach upset of pain (Gastrointestinal disorders) | 513 (513) | 487 (487) | 505 (505) | 495 (495) | 258 (258) | 255 (255) | 247 (247) | 240 (240)
Nausea (Gastrointestinal disorders) | 355 (355) | 346 (346) | 364 (364) | 337 (337) | 182 (182) | 173 (173) | 182 (182) | 164 (164)
Constipation (Gastrointestinal disorders) | 568 (568) | 573 (573) | 547 (547) | 594 (594) | 268 (268) | 300 (300) | 279 (279) | 294 (294)
Diarrhea (Gastrointestinal disorders) | 575 (575) | 600 (600) | 584 (584) | 591 (591) | 286 (286) | 289 (289) | 298 (298) | 302 (302)
Increased burping (Gastrointestinal disorders) | 229 (229) | 251 (251) | 240 (240) | 240 (240) | 109 (109) | 120 (120) | 131 (131) | 120 (120)
Bad taste in mouth (General disorders) | 229 (229) | 231 (231) | 234 (234) | 226 (226) | 120 (120) | 109 (109) | 114 (114) | 117 (117)
Kidney stones (Renal and urinary disorders) | 24 (24) | 25 (25) | 24 (24) | 25 (25) | 12 (12) | 12 (12) | 12 (12) | 13 (13)
Kidney failure or dialysis (Renal and urinary disorders) | 11 (11) | 8 (8) | 9 (9) | 10 (10) | 6 (6) | 5 (5) | 3 (3) | 5 (5)
Skin rash (Skin and subcutaneous tissue disorders) | 352 (352) | 361 (361) | 344 (344) | 369 (369) | 165 (165) | 187 (187) | 179 (179) | 182 (182)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No